CLINICAL TRIAL: NCT01721655
Title: Determining the Effect of Spironolactone on Electrolyte Supplementation in Preterm Infants With Chronic Lung Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West Virginia University Healthcare (Other)
Responsible Party: Principal Investigator, Courtney Brown Sweet, Pediatric Clinical Pharmacy Specialist, West Virginia University Healthcare
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-24305
Record Dates: First submitted 2012-11-01; First posted 2012-11-06 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Lung Disease; Bronchopulmonary Dysplasia
Keywords: Spironolactone; Preterm Infants; Chronic Lung Disease; Bronchopulmonary Dysplasia; Electrolyte Supplementation
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spironolactone (Active Comparator): Oral spironolactone suspension dosed at 3 mg/kg/day will be administered once-daily to the patients assigned to the treatment arm.
  Interventions: Drug: Spironolactone
- Placebo suspension (Placebo Comparator): An oral placebo suspension dosed at 3 mg/kg/day administered once-daily will be given to patients in the placebo arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — Patients will continue to receive standard of care as if they were not enrolled in the study. All patients will receive oral chlorothiazide 40 mg/kg/day divided twice-daily, electrolyte supplementation as needed based on a standard algorithm, and if needed, rescue enteral furosemide 2 mg/kg/day. The intervention will be enteral spironolactone 3 mg/kg once daily
  Other Names: Aldactone
  Arms: Spironolactone
Drug: Placebo — Patients will continue to receive standard of care as if they were not enrolled in the study. All patients will receive oral chlorothiazide 40 mg/kg/day divided twice-daily, electrolyte supplementation as needed based on a standard algorithm, and if needed, rescue enteral furosemide 2 mg/kg/day.
  Other Names: an equivalent placebo
  Arms: Placebo suspension

SUMMARY:
Bronchopulmonary dysplasia (BPD), also known as chronic lung disease (CLD), is a major complication of premature birth and is associated with a significant increased risk of complications including death. Diuretics have been used for decades in babies with BPD and are considered a standard of care. Patients receive electrolyte supplementation to replace the electrolytes removed by the diuretics. Spironolactone is not as good as other diuretics at removing extra fluid, but it is different from chlorothiazide and furosemide because instead of removing potassium, it actually can increase potassium levels in our body. Spironolactone is used with chlorothiazide to try to minimize the potassium lost; therefore, reduce the electrolyte supplementation needed. However, studies have suggested that preterm babies aren´t developed enough to appropriately respond to spironolactone. Also, one study has shown that adding spironolactone to chlorothiazide in patients with BPD has no effect on whether or not patients receive electrolyte supplementation. This study will examine whether there is a difference in the amount of electrolyte supplementation between patients receiving chlorothiazide only or chlorothiazide plus spironolactone. the investigators hypothesize there will be no difference in the amount of electrolyte supplementation between the two groups.

DETAILED DESCRIPTION:
Bronchopulmonary dysplasia (BPD), also known as chronic lung disease (CLD), is a major complication of premature birth and is associated with significant morbidity and mortality. Bronchopulmonary dysplasia most commonly affects preterm infants who have required prolonged aggressive mechanical ventilation and/or oxygen supplementation. Risk factors associated with BPD include degree of prematurity, infection, mechanical ventilation, oxygen concentration, and nutritional status. Despite significant advances in the care of preterm infants and improved survival, the incidence of BPD has been fairly static over the past decade.

Diuretics and fluid restriction are considered a mainstay of therapy in the management of BPD to combat interstitial alveolar edema. Short courses of furosemide followed by long-term therapy using a thiazide diuretic with concurrent spironolactone have shown improvement in pulmonary function and better outcomes. Double-blinded, randomized, placebo-controlled trials have shown improvement in pulmonary compliance, airway resistance, infants alive at discharge, and a decrease in fraction of inspired oxygen and need for furosemide boluses.

Spironolactone is a competitive aldosterone receptor antagonist that acts on the distal convoluted tubule and collecting duct to facilitate sodium excretion while conserving potassium and hydrogen ions. Since only a minimal amount of sodium filtered by the glomerulus reaches the distal tubule, spironolactone is considered a weak diuretic. Spironolactone is primarily used with chlorothiazide for its potassium-sparing effect to reduce the need for electrolyte supplementation. There has only been one prospective, randomized, double-blind, placebo-controlled study comparing chlorothiazide with or without the addition of spironolactone in premature infants with chronic lung disease. This study demonstrated no difference between the groups in the need for electrolyte supplementation, electrolyte balance, or pulmonary function. In addition, preterm infants' distal tubules may respond inadequately to aldosterone; thereby, limiting the role of spironolactone in this patient population.

In the neonatal population, spironolactone is primarily used in addition with chlorothiazide for its potassium-sparing effects to reduce the need for electrolyte supplementation. However, evidence and current practice suggests the majority of patients still receive electrolyte supplementation. One study evaluated spironolactone's effect on the need for electrolyte supplementation, but there is no published data with a primary outcome evaluating spironolactone's effect on the quantity of electrolyte supplementation. We hypothesize there will be no difference in the amount of electrolyte supplementation between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* The attending makes the decision to start enteral chlorothiazide for long-term diuretic therapy.
* Gestational age < 32 weeks at time of delivery
* If patient is currently receiving furosemide and electrolyte supplements, these must be discontinued prior to enrollment.

Exclusion Criteria:

* Renal anomaly
* Receiving maintenance IV fluids for more than the previous 48 hours
* Any contraindication to receiving enteral medication
* Serum Na < 132 mEq/L
* Serum K < 3.0 mEq/L
* Serum Cl < 92 mEq/L
* Presence of ostomy of any sort

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Dose of potassium chloride in milliequivalents/kg/day | Day 28
  The primary objective of this study is to assess the effect of spironolactone on the quantity of electrolyte supplementation in preterm infants receiving a standard regimen for chronic lung disease. The primary endpoint compared between groups will be the dose of potassium chloride in milliequivalents/kg/day from baseline to day 28.

SECONDARY OUTCOMES:
Requirement of electrolyte supplementation | Day 28
  Treatment and control groups will be compared to assess if there is a difference between the need for electrolyte supplementation.
Analyze the use of furosemide rescue doses | Day 28
  The groups will be compared to assess the difference in the need for rescue furosemide doses (enteral furosemide at 2 mg/kg once daily).
Number of furosemide doses utilized | Day 28
  The total number of rescue furosemide doses utilized will be compared between groups.
Escalation in respiratory support | Day 28
  Groups will be compared to determine if there is a difference in the need for an escalation in respiratory support throughout the study period. Escalation in respiratory support is defined as an increase in mean airway pressure for patients on the ventilator, 20% or greater increase in the fraction of inspired oxygen, or an escalation in the mode of support.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney B Sweet, PharmD, Principal Investigator — WVU Healthcare
Locations (1):
- West Virginia University Healthcare, Morgantown, West Virginia, United States

REFERENCES:
- [Background] Jeng SF, Hsu CH, Tsao PN, Chou HC, Lee WT, Kao HA, Hung HY, Chang JH, Chiu NC, Hsieh WS. Bronchopulmonary dysplasia predicts adverse developmental and clinical outcomes in very-low-birthweight infants. Dev Med Child Neurol. 2008 Jan;50(1):51-7. doi: 10.1111/j.1469-8749.2007.02011.x. PMID 18173631
- [Background] Gien J, Kinsella JP. Pathogenesis and treatment of bronchopulmonary dysplasia. Curr Opin Pediatr. 2011 Jun;23(3):305-13. doi: 10.1097/MOP.0b013e328346577f. PMID 21494147
- [Background] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896
- [Background] Smith VC, Zupancic JA, McCormick MC, Croen LA, Greene J, Escobar GJ, Richardson DK. Trends in severe bronchopulmonary dysplasia rates between 1994 and 2002. J Pediatr. 2005 Apr;146(4):469-73. doi: 10.1016/j.jpeds.2004.12.023. PMID 15812448
- [Background] Northway WH Jr, Rosan RC, Porter DY. Pulmonary disease following respirator therapy of hyaline-membrane disease. Bronchopulmonary dysplasia. N Engl J Med. 1967 Feb 16;276(7):357-68. doi: 10.1056/NEJM196702162760701. No abstract available. PMID 5334613
- [Background] Jobe AH, Ikegami M. Mechanisms initiating lung injury in the preterm. Early Hum Dev. 1998 Nov;53(1):81-94. doi: 10.1016/s0378-3782(98)00045-0. PMID 10193929
- [Background] Jobe AJ. The new BPD: an arrest of lung development. Pediatr Res. 1999 Dec;46(6):641-3. doi: 10.1203/00006450-199912000-00007. No abstract available. PMID 10590017
- [Background] Shah PS. Current perspectives on the prevention and management of chronic lung disease in preterm infants. Paediatr Drugs. 2003;5(7):463-80. doi: 10.2165/00128072-200305070-00004. PMID 12837119
- [Background] Tropea K, Christou H. Current pharmacologic approaches for prevention and treatment of bronchopulmonary dysplasia. Int J Pediatr. 2012;2012:598606. doi: 10.1155/2012/598606. Epub 2012 Jan 3. PMID 22262977
- [Background] Biniwale MA, Ehrenkranz RA. The role of nutrition in the prevention and management of bronchopulmonary dysplasia. Semin Perinatol. 2006 Aug;30(4):200-8. doi: 10.1053/j.semperi.2006.05.007. PMID 16860160
- [Background] Albersheim SG, Solimano AJ, Sharma AK, Smyth JA, Rotschild A, Wood BJ, Sheps SB. Randomized, double-blind, controlled trial of long-term diuretic therapy for bronchopulmonary dysplasia. J Pediatr. 1989 Oct;115(4):615-20. doi: 10.1016/s0022-3476(89)80297-5. PMID 2677293
- [Background] Kao LC, Durand DJ, McCrea RC, Birch M, Powers RJ, Nickerson BG. Randomized trial of long-term diuretic therapy for infants with oxygen-dependent bronchopulmonary dysplasia. J Pediatr. 1994 May;124(5 Pt 1):772-81. doi: 10.1016/s0022-3476(05)81373-3. PMID 8176568
- [Background] Kao LC, Warburton D, Cheng MH, Cedeno C, Platzker AC, Keens TG. Effect of oral diuretics on pulmonary mechanics in infants with chronic bronchopulmonary dysplasia: results of a double-blind crossover sequential trial. Pediatrics. 1984 Jul;74(1):37-44. PMID 6377221
- [Background] Engelhardt B, Blalock WA, DonLevy S, Rush M, Hazinski TA. Effect of spironolactone-hydrochlorothiazide on lung function in infants with chronic bronchopulmonary dysplasia. J Pediatr. 1989 Apr;114(4 Pt 1):619-24. doi: 10.1016/s0022-3476(89)80708-5. PMID 2926575
- [Background] Brion LP, Primhak RA, Ambrosio-Perez I. Diuretics acting on the distal renal tubule for preterm infants with (or developing) chronic lung disease. Cochrane Database Syst Rev. 2002;(1):CD001817. doi: 10.1002/14651858.CD001817. PMID 11869608
- [Background] Segar JL. Neonatal diuretic therapy: furosemide, thiazides, and spironolactone. Clin Perinatol. 2012 Mar;39(1):209-20. doi: 10.1016/j.clp.2011.12.007. Epub 2011 Dec 29. PMID 22341547
- [Background] Hoffman DJ, Gerdes JS, Abbasi S. Pulmonary function and electrolyte balance following spironolactone treatment in preterm infants with chronic lung disease: a double-blind, placebo-controlled, randomized trial. J Perinatol. 2000 Jan-Feb;20(1):41-5. doi: 10.1038/sj.jp.7200307. PMID 10693099
- [Background] Sulyok E, Varga F, Gyory E, Jobst K, Csaba IF. Postnatal development of renal sodium handling in premature infants. J Pediatr. 1979 Nov;95(5 Pt 1):787-92. doi: 10.1016/s0022-3476(79)80737-4. PMID 490250
- [Background] Spitzer A. The role of the kidney in sodium homeostasis during maturation. Kidney Int. 1982 Apr;21(4):539-45. doi: 10.1038/ki.1982.60. PMID 7047859